CLINICAL TRIAL: NCT00976534
Title: A Phase IIa Randomised, Double-blind, Placebo Controlled, Parallel Group, Multicentre Study Evaluating the Efficacy, Safety, Tolerability and Pharmacokinetics of AZD1386 After 3 Weeks of Treatment in Patients With Posttraumatic Neuralgia (PTN) and Postherpetic Neuralgia (PHN)
Brief Title: Study to Evaluate Efficacy, Safety, Tolerability and Pharmacokinetics of AZD1386 in Patients With Peripheral Neuropathic Pain
Acronym: AVANT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to results in another study (NCT00878501).
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca Pharmaceuticals, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5090C00018
Record Dates: First submitted 2009-09-09; First posted 2009-09-14 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Pain; Neuropathic Pain
Keywords: Analgesic effect; Peripheral Neuropathic pain; Posttraumatic Neuralgia (PTN); Postherpetic Neuralgia (PHN)
MeSH Terms: conditions — Pain; Neuralgia; Neuralgia, Postherpetic | interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1386
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — 90 mg, capsules, oral, during 3 weeks
  Arms: 1
Drug: Placebo — capsules, oral, during 3 weeks
  Arms: 2

SUMMARY:
The primary aim of this study is to investigate if AZD1386 is efficacious as an analgesic in patients with peripheral neuropathic pain. This will be done by comparing the effect of AZD1386 to placebo ("inactive substance") on pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful symptoms due to neuropathic pain
* Provision of signed informed consent
* Non pregnant females

Exclusion Criteria:

* Other pain conditions that may confound assessment of neuropathic pain, as judged by the investigator
* History, and/or presence of somatic disease, which may interfere with the objectives of the study as judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-09; Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NRS pain (12 h-recall) | Morning and evening 12 hour recall

SECONDARY OUTCOMES:
Response rate, defined as any of the following:NRS (12 h recall) reduced by 30% compared to baseline and NRS (12 h recall) reduced by 50% compared to baseline | Morning and evening 12 hour recall
Response rate, defined as any of the following: At least "much improved" on Patient Global Impression of Change global and at least "much improved" on PGIC pain | Day 8, 15 and 22
Response rate, defined as any of the following: Change from baseline in Brief Pain Inventory Short Form and Change from baseline in Pain Quality Assessment Scale | Day 1 and 22

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Leff, md, Study Director — AstraZeneca R&D Wilmington, USA; Rolf Karlsten, MD, Study Chair — AstraZeneca R&D Södertälje, Sweden
Locations (12):
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Toronto, Ontario
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Arhus C
- France (3):
  - Research Site, Boulogne-Billancourt
  - Research Site, Clermont-Ferrand
  - Research Site, Nice
- United Kingdom (4):
  - Research Site, Bradford
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester